CLINICAL TRIAL: NCT04863521
Title: Pilot MHP 3.0 in Two Clinical Settings to Evaluate Acceptability and Feasibility of MHP
Brief Title: Evaluation of MHP 3.0 in Two Clinical Settings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Naima Health LLC (Other)
Collaborators: University of Pittsburgh (Other); Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDC-PHASEII-003
Record Dates: First submitted 2021-04-16; First posted 2021-04-28 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Telemedicine

STUDY DESIGN:
Intervention Model Description: Users recruited at Obstetrix Medical Group of Houston will participate in a pilot study that includes facilitating access to the app and will be followed throughout their pregnancy using online surveys. Users at the UPMC Healthcare System are already using the app as part of their routine care and will be asked to complete an online survey about their user experience.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHP Users (Experimental): A subset of the population within the clinical setting will be requested to participate in this pilot while the rest of the population will receive standard of care.
  Interventions: Other: MHP

INTERVENTIONS:
Other: MHP — MyHealthyPregnancy app (MHP 3.0) is a mHealth app specifically focused on detection and referral for depression and IPV (Intimate Partner Violence) risk, in addition to its other pregnancy risk detection and support features.

SUMMARY:
The purpose of this study is to assess the acceptability and feasibility of the use of MyHealthyPregnancy (MHP) 3.0 in clinical practice over a 1 year period of time. The investigators will pilot MHP 3.0 (Spanish and English language options) at practice sites at the Obstetrix Medical Group of Houston, Texas and the UPMC (University of Pittsburgh Medical Center) Healthcare System. Patient and care team feedback will be assessed throughout this study. Patients at Obstetrix Medical Group of Houston will be assessed using 4 short acceptability and feasibility surveys administered by the Naima Health team using a link for an online survey during the study term: at baseline, week 14-18, week 24-28, and week 34-36. A subset of participants at UPMC will also be asked to complete user surveys.

DETAILED DESCRIPTION:
For this study the investigators pilot MHP products in two clinical settings to determine their acceptability and feasibility in clinical practice. The investigators will pilot MHP 3.0 (Spanish and English language options) at practice sites at the Obstetrix Medical Group of Houston, Texas and the UPMC Healthcare System. Participants will receive MHP to use as part of their prenatal care, along with communication from the prescribing provider about how the app will be used and when the provider will have access to their information.

Population and Sample Size: The investigators will recruit a sample of 75 patients from the Obstetrix Medical Group clinical sites in women's first trimester of pregnancy. The investigators will over sample for Spanish speakers (approximately 20% of our population). Women will be eligible for recruitment if they are at least 18 years old, are currently pregnant and under the care of a participating provider/clinic, own a smartphone, and are literate in English or Spanish. We will recruit 75 patients patients who are currently using MHP as part of their routine care at the UPMC Healthcare system to complete a user online survey to discuss their experience with the app.

At Obstetrix Medical Group of Houston, recruitment staff will identify eligible women to match our demographic requirements, introduce the study during an initial prenatal appointment, and then consent women to the study.

Data sources and collection:

Patients at Obstetrix Medical Group of Houston: A short acceptability and feasibility survey will be administered by the Naima Health team online four times during the study term. A final interview will be conducted by phone between weeks 36-42 with a sample of 10 - 15 study participants.

Patients at UPMC Healthcare system: Patients who have been prescribed the app as part of their routine care will be invited to participate in an online survey.

Analytic Plan and Sample Size Considerations:

The investigators will focus on feasibility (a priori defined as ≥ 67% completion of weekly questionnaires administered through the app) and acceptability (a priori defined as satisfaction scores of ≥ 4 on a 7-point Likert scale among ≥80% participants) as primary outcomes for this aim. Descriptive statistics will be used to characterize baseline demographic characteristics of the participants. The investigators will use point estimates (i.e. means and sample proportions) and 95% confidence intervals to characterize the sample with respect to baseline demographic characteristics. Debriefing interview transcripts will be coded for themes of acceptability, satisfaction, and barriers to app use.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age
* Currently pregnant and in gestational week 12 or less
* Is under the care of a participating provider/clinic
* Owns a smartphone
* Spanish or English native speaker

Exclusion Criteria:

* Under 18 years of age
* Not pregnant at time of enrollment
* Is pregnant but over 12 weeks of gestational age
* Provider is not part of the study
* Does not own a smartphone
* Native language is not Spanish or English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be pregnant
Enrollment: 150 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of patients that screen positive | 8 months
  Measured by the number of patients who screen positive for depression and/or intimate partner violence through the app compared to the number of patients who have screened positive for depression and/or intimate partner violence historically through routine prenatal care. Higher numbers mean better outcomes.
Percentage of questionnaires completed | 8 months
  Measured by calculating the percentage of questionnaires completed by each user from the total administered through the MHP app. Values would range from 0% to 100%. Higher numbers mean better outcomes.
Usability Questionnaire | 8 months
  This questionnaire will assess subjective opinions about the usability of MHP. This questionnaire includes 7 questions that will use a Likert scale anchored from 1/strongly disagree to 5/strongly agree. The minimum value is 7 and the maximum value of 35. Higher numbers mean better outcomes.
Acceptability Questionnaire | 8 months
  This questionnaire will assess subjective opinions about the acceptability of the content in MHP. This questionnaire includes 6 questions that will use a Likert scale anchored from 1/strongly disagree to 5/strongly agree. The minimum value is 6 and the maximum value of 30. Higher numbers mean better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrix Medical Center Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No